CLINICAL TRIAL: NCT07338643
Title: The Auxiliary Effect of Artificial Intelligence in the Detection of Precancerous Lesions in Proximal Colon Cancer: A Multicenter Randomized Controlled Study
Brief Title: The Auxiliary Effect of Artificial Intelligence in the Detection of Precancerous Lesions in Proximal Colon Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Limian Er (Other)
Responsible Party: Sponsor-Investigator, Limian Er, The director of the Endoscopy Department of the Fourth Hospital of Hebei Medical University, Hebei Medical University Fourth Hospital
Organization: Hebei Medical University Fourth Hospital (Other)
Other Study IDs: 2025KS177
Record Dates: First submitted 2025-12-18; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Abdominal Pain; Black Stools; Constipation; Diarrhea
MeSH Terms: conditions — Abdominal Pain; Melena; Constipation; Diarrhea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- AI group
  Interventions: Procedure: AI group
- Series group
  Interventions: Procedure: Serial group
- Standard group
  Interventions: Procedure: Standard colonoscopy group

INTERVENTIONS:
Procedure: AI group — Full AI assistance was used throughout the standard colonoscopy procedure.
  Groups: AI group
Procedure: Serial group — After normal withdrawal of the colonoscope to the splenic flexure during standard colonoscopy, full AI assistance was initiated. The colonoscope was re-entered to the ileocecal region for observation. Any missed lesions were recorded.
  Groups: Series group
Procedure: Standard colonoscopy group — The standard colonoscopy procedure was performed as usual
  Groups: Standard group

SUMMARY:
The investigators conducted a multicenter randomized controlled trial to explore the adjuvant effect of artificial intelligence in the detection of precancerous lesions in the proximal colon.This is a prospective, multicenter, single-blind, parallel randomized controlled trial.During the colonoscopy retraction process, the investigators aimed to compare the detection rates of proximal colon adenomas with and without the assistance of an AI(Artificial Intelligence) diagnostic device.

ELIGIBILITY:
Inclusion Criteria:

1.Patients with symptoms such as abdominal pain, black stools, constipation, or diarrhea undergo colonoscopy for diagnostic purposes.

Exclusion Criteria:

1. Those with inflammatory bowel disease, colorectal cancer and surgical history, as well as those with familial polyposis syndrome
2. Those with intestinal obstruction or malignant tumors
3. Patients with colorectal lesions that need to be treated in stages.
4. Other contraindications for colonoscopy examination.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with symptoms such as abdominal pain, black stools, constipation, or diarrhea
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2026-02-26 (Estimated); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Adenoma detection rate | Day 1
  The proportion of patients who have at least one adenoma detected during colonoscopy examination
Average adenoma detection rate | Day 1
  The result is the number of adenomas detected by colonoscopy divided by the total number of colonoscopies performed.

CONTACTS AND LOCATIONS:
Overall Officials: Li mian Er, Study Director — Hebei Medical University Fourth Hospital
Locations (1):
- the Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

REFERENCES:
- [Background] Luo Y, Zhang Y, Liu M, Lai Y, Liu P, Wang Z, Xing T, Huang Y, Li Y, Li A, Wang Y, Luo X, Liu S, Han Z. Artificial Intelligence-Assisted Colonoscopy for Detection of Colon Polyps: a Prospective, Randomized Cohort Study. J Gastrointest Surg. 2021 Aug;25(8):2011-2018. doi: 10.1007/s11605-020-04802-4. Epub 2020 Sep 23. PMID 32968933
- [Background] Wu J, Zhang Q, Li X, Bai T, Hou X, Li G, Song J. The Effect of the Second Forward View on the Detection Rate of Sessile Serrated Lesions in the Proximal Colon: A Single-Center Prospective Randomized Controlled Study. Clin Transl Gastroenterol. 2025 Feb 1;16(2):e00805. doi: 10.14309/ctg.0000000000000805. PMID 39688959
- [Background] Leggett B, Whitehall V. Role of the serrated pathway in colorectal cancer pathogenesis. Gastroenterology. 2010 Jun;138(6):2088-100. doi: 10.1053/j.gastro.2009.12.066. PMID 20420948
- [Background] Kim HY, Kim SM, Seo JH, Park EH, Kim N, Lee DH. Age-specific prevalence of serrated lesions and their subtypes by screening colonoscopy: a retrospective study. BMC Gastroenterol. 2014 Apr 28;14:82. doi: 10.1186/1471-230X-14-82. PMID 24775268
- [Background] Huang J, Chan PSF, Pang TWY, Choi P, Chen X, Lok V, Zheng ZJ, Wong MCS. Rate of detection of serrated lesions at colonoscopy in an average-risk population: a meta-analysis of 129,001 individuals. Endosc Int Open. 2021 Mar;9(3):E472-E481. doi: 10.1055/a-1333-1776. Epub 2021 Feb 19. PMID 33655052
- [Background] 王人杰, 张晓兰, 蔡继东, 等. 结直肠息肉的规范化诊疗[J]. 中华胃肠外科杂志, 2024, 27(6): 583-590.
- [Background] 叶倩云,刘凤斌.大肠息肉发病相关风险因素及方法学研究[J].中华中医药杂志, 2018,33(3):4. DOI:CNKI:SUN:BXYY. 0.2018-03-080.